CLINICAL TRIAL: NCT05149885
Title: A Feasibility Study of a Non-Invasive Wearable Device in Assessing Airway Responsiveness Related Parameters During Methacholine Challenge Test (MCT)
Brief Title: A Feasibility Study of SenseGuard to Assess Airway Responsiveness During Methacholine Challenge Test (MCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NanoVation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PD-CLN-001
Record Dates: First submitted 2021-11-03; First posted 2021-12-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational SenseGuard Device (Experimental): Subjects with suspected diagnosis of Asthma and eligible for MCT will be recruited to the study.
  The MCT procedure will be performed as usual, with the addition of SG measurements after each spirometry for each Methacholine dose.
  Interventions: Device: SenseGuard monitoring

INTERVENTIONS:
Device: SenseGuard monitoring — All subjects that recruited to the study will undergo MCT as usual with the addition of SG measurement after each Methacholine dose and spirometry test.

SUMMARY:
SenseGuard (SG) is an innovative device for respiratory monitoring. At this study SG measurement will be integrated in a Methacholine Challenge Test (MCT) for monitoring changes in airway obstruction occurred during MCT in parallel to spirometry.

DETAILED DESCRIPTION:
SenseGuard (SG) is a wireless wearable medical device intended for monitoring of patient's breathing. It allows to seamlessly monitor patient's tidal breathing, at rest or during daily activities, and to extract critical respiratory parameters, such as respiration rate (RR) and durations, ratios and variability of phases within the breath-cycle, including: inspired breath (Ti) and expired breath (Te).

The study goal is to evaluate the capability of SG to measure clinical changes in respiratory parameters.

During Methacholine Challenge Test (MCT), asthma patients demonstrate airway responsiveness due to airway obstruction. SG will be used to measure respiratory parameters during MCT in parallel to spirometry and the correlation between measurable respiratory parameters will be assessed.

Successful study results will demonstrate the capability of SG to measure changes in airway obstruction leading to future implementation of SG for monitoring of patients with respiratory diseases and improvement of their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18.
* Eligible for MCT procedure. The contradictions to MCT are listed as exclusion criteria.
* Provision of a signed and dated informed consent form.
* Subject who receives one of the following medications, that decrease bronchial hyperresponsiveness, is required for a washout period, before conducting the MCT: inhaled bronchodilators, oral albuterol , inhaled and oral glucocorticoids, leukotriene modifying agents, theophylline, cromolyn, and anti-histamines due to their anticholinergic effect.

Exclusion Criteria:

* Subjects who have known contradictions to MCT, including:

  * Tolerate inhalation of the challenge agents
  * Low baseline FEV1: Airflow limitations in FEV1 less than 60% predicted or 1.5L (baseline FEV1 of < 1.5 L or < 60% predicted).
  * Spirometry quality: inability to consistently reproduce quality spirometry
  * Cardiovascular problems: recent myocardial infarction within past three months, uncontrolled hypertension, known aortic aneurysm
  * Recent ophthalmologic surgery or patients at risk for intracranial pressure elevation.
  * Pregnancy and nursing mothers: Methacholine is a pregnancy category C drug and it is not known whether it is excreted in breast milk or is associated with fetal abnormalities. Women subjects will be asked to sign a statement, as part of the Informe Consent Form, that they are not pregnant or nursing mothers).
* Inability to provide informed consent.
* Known allergic reactions to materials used in the components of the SG, i.e., polyethylene or silicon, or gold, nickel, copper or alloys containing any of the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Respiratory parameters (Inhalation and Exhalation time and ratio) measured by SG during MCT can indicate for changes in airway obstruction occurred in positive MCT | 6 months
  SG respiratory parameters(Inhalation and Exhalation (I/E) time and ratio), can measure successfully changes in respiratory parameters during MCT procedure, in at least of 70% of the subjects with MCT positive result (FEV1 < 20% of predicted FEV1).

SECONDARY OUTCOMES:
SG respiratory parameters (Inhalation and Exhalation time and ratio) are in correlation with Spirometry values (FEV1) obtained during MCT | 6 months
  There is at least 70% correlation between changes in respiratory parameters measured by SG (Inhalation and Exhalation (I/E) time and ratio),and by Spirometry values (%FEV1 reduced from baseline) for at least 70% of subjects participating in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Nicosia Lung Center, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months